CLINICAL TRIAL: NCT01456013
Title: A Study to Evaluate RenalGuard® System Safety & Efficacy When Compared With Standard Care in the Prevention of Contrast Induced NephRopathy in the SettinG of a Catheterization Laboratory
Brief Title: Evaluation of RenalGuard® System to Reduce the Incidence of Contrast Induced Nephropathy in At-Risk Patients
Acronym: CIN-RG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CardioRenal Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RGS001D
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Contrast Induced Nephropathy
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Therapy (Active Comparator): Standard of care for patients at risk of CIN
  Interventions: Drug: Standard Therapy
- RenalGuard Therapy (Experimental): Induced Diuresis with Matched Replacement
  Interventions: Device: RenalGuard Therapy

INTERVENTIONS:
Device: RenalGuard Therapy — Induced Diuresis with matched replacement
  Arms: RenalGuard Therapy
Drug: Standard Therapy — Standard of care for patients at risk of CIN
  Arms: Standard Therapy

SUMMARY:
Contrast-Induced Nephropathy (CIN) can occur when patients with pre-existing kidney problems undergo procedures that use iodinated contrast media, such as cardiac catheterizations. RenalGuard Therapy was developed to enable the patient to clear the contrast out of their kidney before it can do significant damage. This study aims to enroll patients with increased risk of developing CIN who are scheduled for a cardiovascular catheterization. Patients will be randomized to either RenalGuard therapy or standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female equal or greater than the age of 18 years old and is able to provide informed consent.
* Subject is scheduled to undergo an elective catheterization procedure
* Hemodynamically stable
* At increased risk of developing CIN
* Subject has agreed to all follow-up testing.

Exclusion Criteria:

* Class 4 Congestive Heart Failure (CHF)or a documented left ventricular ejection fraction < 30%
* Is anuric or has undergone renal replacement therapy within the past month, or has a known inability to have a Foley catheter placed.
* Subject has been hospitalized or treated medically for any change in renal function over the past week (i.e. dialysis, etc.), or a significant change in renal function is noted at time of screening.
* Has documented severe Aortic Stenosis.(Note: Subjects who have undergone successful replacement or repair of their aortic valve are not excluded.)
* Currently has a known clinically significant electrolyte imbalance or clinically significant arrhythmias which compromise subject's hemodynamic state.
* Patient has severe anemia (hemoglobin < 8.0 g/dL) at screening
* Has received contrast within 10 days of procedure or has a planned additional cardiac or renal or other major surgical procedure within the 7 day follow-up period.
* Has ruled in for a Serious Heart Attack within 48 hours of the planned procedure
* Has documented respiratory insufficiency as evidenced by an oxygen saturation of < 90% on room air assessed on day of procedure.
* Planned addition, discontinuation or dose adjustment of nephrotoxic drugs
* Subject has a known hypersensitivity to furosemide and/or the contrast agent being used.
* Subject is currently, plans, or has been enrolled in another clinical study involving use of an investigational drug or device within the prior 30 days.
* Subject is pregnant or breastfeeding.
* Subject is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2012-01; Primary Completion 2018-03 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Contrast Induced Nephropathy | 72 hours

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 90 days
Mean peak increase in serum creatinine post contrast administration | 72 hours
Proportion of patients who develop CIN at 7 days post contrast administration | 7 days
Proportion of patients who maintain a rise in serum creatinine at 7 days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Davidson, MD, Principal Investigator — Northwestern University; Richard Solomon, MD, Principal Investigator — University of Vermont; Roxana Mehran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (30):
- United States (30):
  - University of Alabama, Birmingham, Alabama
  - Torrance Medical Center, Torrance, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Clearwater Cardiovascular, Clearwater, Florida
  - University of Florida, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Advocate Good Samaritan, Downers Grove, Illinois
  - Advocate Health, Naperville, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - St. Elizabeth's Hospital, Brighton, Massachusetts
  - Cape Cod Healthcare, Hyannis, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Northern Michigan Hospital, Petoskey, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Joseph Medical Center, Saint Charles, Missouri
  - NYU Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - Montefiore Medical Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Rex Hospital, Raleigh, North Carolina
  - St. John Research Institute, Bartlesville, Oklahoma
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Guthrie Medical Center, Sayre, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Austin Heart Central, Austin, Texas
  - Baylor Scott & White, Plano, Texas
  - Austin Heart Round Rock, Round Rock, Texas